CLINICAL TRIAL: NCT02707822
Title: The Influence of ABCB1、CYP3A4、CYP3A5、POR Genetic Polymorphism and Other Factors on Tacrolimus Blood Concentration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201512005RINC
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Transplantation; Liver Transplantation
Keywords: tacrolimus; pharmacokinetics; gene polymorphism; clinical factors

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- kidney or liver transplantation: Renal or liver transplant recipients with tacrolimus as immunosuppressive drugs.
  Interventions: Other: Clinical and genetic factors

INTERVENTIONS:
Other: Clinical and genetic factors

SUMMARY:
The purpose of the study is to identify factors that may influence tacrolimus (TAC) pharmacokinetics, and the impact of gene polymorphism (ABCB1, CYP3A4, CYP3A5, POR) on pharmacokinetics of TAC in Taiwanese.

DETAILED DESCRIPTION:
TAC is one of the most important immunosuppressive agents for organ transplantation. In some patients the dose and concentration of TAC are difficult to adjust because of its narrow therapeutic index and variable pharmacokinetics.

Many factors affect the pharmacokinetics of TAC. Literature suggests that ABCB1, CYP3A4, CYP3A5, POR gene polymorphisms may affect the pharmacokinetics of TAC. In addition, the distribution of TAC is affected by hematocrit and albumin concentrations. The pharmacokinetics of TAC may also be affected by total protein, total bilirubin, creatinine, AST, ALT, gender, age, drug interactions, and so on.

This study intends to analyze the influence of various factors, including drugs, on the pharmacokinetics of TAC.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplants or liver transplants
* 20 - 65 years old
* receiving tacrolimus as immunosuppressive drugs

Exclusion Criteria:

* Human immunodeficiency virus-positive status
* Retransplantation or multiorgan transplantation
* non-Asian

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal or liver transplant recipients who underwent transplantation at National Taiwan University Hospital, and were treated with tacrolimus.
Sampling Method: Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Dose-normalized tacrolimus concentration | Within the first 6 months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Kun Tsai, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan